CLINICAL TRIAL: NCT01279642
Title: The Use of Doppler Vascular Ultrasound by Nurses During the Placement of Peripherally Inserted Central Venous Catheters in Children: Clinical, Randomized and Controlled Trial.
Brief Title: Placement of Peripherally Inserted Central Venous Catheters (PICC) in Children Guided by Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Mavilde LG Pedreira, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1967/06; CNPq Grant nº. 476295/2004-1. (Other: National Council Scientific Development Brazil)
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2010-07

CONDITIONS: Cardiovascular Infections; Peripheral Vascular Disease
Keywords: Catheterization, Peripheral; Ultrasonography, Interventional; Nursing; Pediatric
MeSH Terms: conditions — Cardiovascular Infections; Peripheral Vascular Diseases | interventions — Ultrasonography; Ultrasonography, Interventional; Vascular Access Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ultrasound (Experimental): Use of ultrasound to PICC placement
  Interventions: Device: ultrasound
- Control group (Active Comparator): PICC placement by inspection and visualization of site
  Interventions: Other: traditional puncture

INTERVENTIONS:
Device: ultrasound — Doppler vascular ultrasound guidance to PICC insertion in children -
  Other Names: vascular doppler ultrasound; interventional ultrasound; vascualr access
  Arms: ultrasound
Other: traditional puncture — traditional approach of PICC insertion by visualization and inspection of insertion site
  Other Names: vascular access
  Arms: Control group

SUMMARY:
Aimed to compare the success in the peripheral intravenous puncture (PIP), progression and placement of PICC in children, according to the use of Doppler vascular ultrasound (DVUS) or traditional method; to identify the influence of the DUVS in the time expended to PICC placement. Methods: Clinical, randomized and controlled trial conducted after ethical merits of research endorsement and the obtaining of consent for those responsible for the children. The sample, calculated in 42 PICC to obtain a power of 0,85, was distributed randomly into two groups, experimental group (EG) and controlled group (CG). To the statistical analyzes Pearson Chi-square, Fisher's Exact Tests, Generalization of Fischer's Exact and Mann-Whitney tests was applied (5%). Of the 42 catheters, 21 (50.0%) were implemented in EG and 21 (50.0%) in CG. The PIP was obtained in the first attempt in 90.5% of the punctures of the EG and in 47.6% of the GC, (p=0.003). PICC were implanted successfully in 18 (85.7%) children of GE and 11 (61.1%) of CG (p = 0.019). The median of the time spent to the procedure was significantly higher (p=0.001) in CG (50 minutes) when compared to EG (median 20 minutes).

DETAILED DESCRIPTION:
Introduction: Peripherally inserted central venous catheters (PICC) are increasingly being used to intravenous therapy in a wide variety of adults and pediatrics patients. Children may have characteristics that could compromise the assertiveness during the catheter placement, even for the more experienced and qualified professionals. In order to search for methods that could lead to the nursing practice innovation seeking for better results in the placement of PICC, this study was designed to analyze the use of Doppler vascular ultrasound (DVUS) to PICC insertion performed by nurses. Objective: To compare the success in the peripheral intravenous puncture (PIP), progression and placement of PICC in children, according to the use of DVUS or traditional method; to identify the influence of the DUVS in the time expended to the placement of PICC in children. Methods: Clinical, randomized and controlled trial conducted in a pediatric surgery ward of a university hospital, from August 17th, 2007 to August 19th, 2008, after ethical merits of research endorsement and the obtaining of consent for those responsible for the children. The sample, calculated in 42 PICC to obtain a power of 0,85, was distributed randomly into two groups, experimental group (EG) and controlled group (CG). The dependent variables were: the success in the PIP, catheter progression and placement. Variables related to children and IV therapy was investigated. To the statistical analyzes Pearson Chi-square, Fisher's Exact Tests, Generalization of Fischer's Exact and Mann-Whitney tests was applied (significance level of 5%). Results: Of the 42 catheters, 21 (50.0%) were implemented in EG and 21 (50.0%) in CG. The PIP was obtained in the first attempt in 90.5% of the punctures of the EG and in 47.6% of the GC, (p=0.003)and the punctures were accomplished to catheter insertion, despite the number of attempts in 76.5% of EG and 41.7% in GC (p = 0.001). The successful to PICC progression was marginally significant result (p=0.069), 69.2% in EG and 44.0% in CG. PICC were implanted successfully in 18 (85.7%) children of GE and 11 (61.1%) of CG (p = 0.019). The median of the time spent to the procedure was significantly higher (p=0.001) in CG (50 minutes) when compared to EG (median 20 minutes). Conclusion: The results obtained lead to the conclusion that the use of USVD to the implementation of the PICC in children promoted greater success in the PIP and in PICC placement, reducing of the time spent to the procedure, but no significant influence was observed regarding the catheter progression.

ELIGIBILITY:
Inclusion Criteria:

* Children in IV Therapy for 7 days or more;
* Peripheral venous vessels indicated to PICC

Exclusion Criteria:

* Patient or family refuse to consent in PICC insertion.
* Patient or family refuse to participate in the research.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Success in PICC placement. | 1 year
  The PICC was placed in the first attempt in 90.5% of the punctures of the ultrasound group and in 47.6% of the control group (p=0.003

SECONDARY OUTCOMES:
Time spent to PICC placement | 1 year
  The median time spent to the procedure was significantly higher (p=0.001) in control group (50 minutes) when compared to ultrasound group (median 20 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Mavilde LG Pedreira, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil